CLINICAL TRIAL: NCT01969357
Title: A Multicenter Randomized, Double-blind, Placebo and Positive Controlled ,Parallel Group ,Phase II Study to Access the Efficacy and Safety of SP2086 Treated Type 2 Diabetes Patients
Brief Title: A Study of the Effectiveness and Safety of SP2086 to Treat Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-SP-201
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: Sp2086; Phase II; monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 50 mg SP2086 (Experimental)
  Interventions: Drug: 50 mg SP2086
- 100 mg SP2086 (Experimental)
  Interventions: Drug: 100 mg SP2086
- 200 mg SP2086 (Experimental)
  Interventions: Drug: 200 mg SP2086
- 100 mg Sitagliptin (Active Comparator)
  Interventions: Drug: 100 mg Sitagliptin

INTERVENTIONS:
Drug: Placebo — Tablets(n=4),once daily for 84 days
  Arms: Placebo
Drug: 50 mg SP2086 — Tablets(n=1),50mg strength+tablets(n=3) 0 mg once daily for 84 days
  Arms: 50 mg SP2086
Drug: 100 mg SP2086 — Tablets(n=1),100 mg strength+tablets(n=3) once 0 mg daily for 84 days
  Arms: 100 mg SP2086
Drug: 200 mg SP2086 — Tablets(n=2),100 mg strength+tablets(n=2) 0mg once daily for 84 days
  Arms: 200 mg SP2086
Drug: 100 mg Sitagliptin — Tablets(n=1),100 mg strength+tablets(n=3),0 mg strength once daily for 84 days
  Arms: 100 mg Sitagliptin

SUMMARY:
SP2086 is a new dipeptidy1 peptidase(DPP)-4 inhibitors. This study aims to explore the effective dose range of SP2086 in Patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 20 Years to 70 Years ,Male and Female diagnosed with type 2 diabetes mellitus
* Patients not on an oral antihyperglycemic agent (OHA) with 7.0% ≤HbA1C ≤10.5%,or not on an OHA for 3 months with 7.0% ≤HbA1C ≤10.5%
* BMI 19~35 kg/m2

Exclusion Criteria:

* Patient has history of type 1 diabetes mellitus
* Patient has history of ketoacidosis
* Patient has history of severe unconscious hypoglycemosis
* Patient has history of acute and chronic pancreatitis or pancreatic injury that may lead to high risk of pancreatitis
* Patient has history of decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistence and clinical
* Patient has history of a history of hypertension, and after antihypertensive treatment, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg
* Patient has severe liver or kidney disease,alanine aminotransferase >2×UNL, Aspartate Aminotransferase >2×upper normal limit(UNL)；total bilirubin >2×UNL； creatinine>1.5 mg/dL (Male,132.6μmol/L) ，>1.4 mg/dL(Female，123.8μmol/L)
* Patient has severe chronic gastrointestinal disease or therapy that may affect drug absorption, such as gastrointestinal surgery
* Patient has severe haematological diseases or other diseases leading to hemolyze and red blood cell unstable (malaria、haemolytic anaemia eg. )
* Patient has other endocrine diseases, for example hyperthyroidism、hypothyroidism、hypercortisolism、multiple endocrine neoplasia and so on
* Patient has history of malignancy
* Patient has history of alcohol or drug abuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
the change from baseline in HbA1c at 12 week | baseline, week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving Less Than (<) 6.5% or <7% HbA1c Levels | week 12
Change From Baseline in Fasting Plasma Glucose at Week 4, 8 and 12 | Baseline, Week 4, 8, 12
Post-meal total and incremental glucose,insulin and C-peptide area under the curve at week 4 ,12 | baseline, week 4 ,12
Change from baseline in Homeostasis model assessment-beta(HOMA-β) at week 4,week12 | baseline, week 4,12week
Change From Baseline in lipid at Week 4, 8 and 12 | baseline, week 4, 8, 12
Change From Baseline in Body Weight at Week 4,8,12 | baseline, Week 4, 8,12

CONTACTS AND LOCATIONS:
Overall Officials: Changyu Pan, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China